CLINICAL TRIAL: NCT02074046
Title: Study of Cancer Stem Cell Vaccine That as a Specific Antigen in Metastatic Adenocarcinoma of the Pancreas
Brief Title: Safety Study of Cancer Stem Cell Vaccine to Treat Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLP-001; 201401 (Other Grant/Funding Number: The research fund of Fuda cancer hospital in Guangzhou)
Record Dates: First submitted 2014-02-25; First posted 2014-02-28 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2014-02

CONDITIONS: Neoplasms, Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- non-cancer stem cell vaccine (Placebo Comparator): The using dosage,frequency and duration of cancer stem cell vaccine are still undetermined.
  Interventions: Biological: cancer stem cell vaccine
- giving low dose vaccine (Experimental): The using dosage,frequency and duration of cancer stem cell vaccine are still undetermined.
  Interventions: Biological: cancer stem cell vaccine
- giving middle dose vaccine (Experimental): The using dosage,frequency and duration of cancer stem cell vaccine are still undetermined.
  Interventions: Biological: cancer stem cell vaccine
- giving high dose vaccine (Experimental): The using dosage,frequency and duration of cancer stem cell vaccine are still undetermined.
  Interventions: Biological: cancer stem cell vaccine

INTERVENTIONS:
Biological: cancer stem cell vaccine

SUMMARY:
Most studies of cancer stem cells (CSC) involve the inoculation of cells from human tumors into immunosuppressed mice, preventing an assessment on the immunologic interactions and effects of CSCs. In this study, the investigators examined the vaccination effects produced by CSC-enriched populations from histologically distinct murine tumors after their inoculation into different syngeneic immunocompetent hosts. Enriched CSCs were immunogenic and more effective as an antigen source than unselected tumor cells in inducing protective antitumor immunity.Immune sera from CSC-vaccinated hosts contained high levels of IgG which bound to CSCs, resulting in CSC lysis in the presence of complement.CTLs generated from peripheral blood mononuclear cells or splenocytes harvested from CSC-vaccinated hosts were capable of killing CSCs in vitro. Mechanistic investigations established that CSC-primed antibodies and T cells were capable of selective targeting CSCs and conferring antitumor immunity.

DETAILED DESCRIPTION:
To assess the feasibility of generating CSC-loaded DC vaccines for clinical use, the investigators will harvest peripheral blood and tumor specimen from patients with Pancreatic Cancer. The investigators will purify T, B cells and generate DCs from the PBMCs of the Pancreatic Cancer patient.On the other hand, investigators will isolate ALDHhigh and ALDHlow tumor cells from the tumor specimen of the Pancreatic Cancer patient using a similar protocol as investigators reported .

Aim 1: To demonstrate, in vitro, the relative cellular anti-Pancreatic Cancer CSC immunity induced by Pancreatic Cancer CSC-DC primed cytotoxic T cells.

Aim 2: To determine, in vitro, specific binding and lysis of Pancreatic Cancer CSCs by antibodies produced by purified B cells from PBMCs stimulated with Pancreatic Cancer CSC-DC.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients must have histologically or cytologically confirmed adenocarcinoma of the pancreas. The site of the primary lesion should be confirmed endoscopically, radiologically, or surgically to be in the pancreas.

  2. Patients must be deemed unresectable due to involvement of critical vasculature, adjacent organ invasion, presence of metastasis, or other medical condition making surgical resection unfavorable.

  3. Patients must have a primary or metastatic lesion measurable in at least one dimension by RECIST criteria within 4 weeks prior to entry of study .

  4. More than 4 weeks must have elapsed from the time of major surgery or completion of the last dose of chemotherapy, radiation therapy, investigational therapy and patients must adequately recover from these effects.

  5. Life expectancy of >3 months. 6. Karnofsky performance status >70%. 7. The patient shows normal organ function according to the following parameters(as measured within six weeks prior to treatment allocation):
* Hemoglobin: Within normal range according to institutional standards;
* Absolute leukocyte count: Within normal range according to institutional standards;
* Absolute lymphocyte count: Within normal range according to institutional standards;
* Platelet count: Within normal range according to institutional standards;
* Alanine aminotransferase: ≤ 2.5 x Upper Limit of Normal (ULN);
* Aspartate aminotransferase: ≤ 2.5 x ULN;
* Total bilirubin: ≤ 1.5 x ULN. In the case of known Gilbert's syndrome ≤ 2 x ULN;
* Serum creatinine: 1.5 x ULN;
* Calculated creatinine clearance: > 50 mL/min . 8. Age >18 years. 9. No history of autoimmune diseases. 10. Ability to understand the study protocol and a willingness to sign a written informed consent document.

Exclusion Criteria:

- 1. Patients receiving anticoagulation therapy. 2. Patients who have received prior gemcitabine or radiation therapy to the pancreatic bed 3. Patients receiving any other investigational agents. 4. Patients with known brain metastases will be excluded because of their poor prognosis and because they often develop progressive neurological dysfunction that would confound the evaluation of neurological and other adverse effects.

5. Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements.

6. Patients who test positive for Hepatitis B virus, Hepatitis C virus or HIV. 7. level 3 hypertension; 8. severe coronary disease; 9. myelosuppression; 10. respiratory disease; 11. brain metastasis; 12. chronic infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The primary study purpose to determine the safety of immunization with cancer stem cells vaccine by the number of participants with adverse events | up to 3 months

SECONDARY OUTCOMES:
The secondary objectives are to evaluate vaccine immune responses to the immunizations by the data of body measurements | 1 month

OTHER OUTCOMES:
The dose of CSC vaccine | up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Biological treatment center in Fuda cancer hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Ning N, Pan Q, Zheng F, Teitz-Tennenbaum S, Egenti M, Yet J, Li M, Ginestier C, Wicha MS, Moyer JS, Prince ME, Xu Y, Zhang XL, Huang S, Chang AE, Li Q. Cancer stem cell vaccination confers significant antitumor immunity. Cancer Res. 2012 Apr 1;72(7):1853-64. doi: 10.1158/0008-5472.CAN-11-1400. PMID 22473314
- See also: Related Info — http://www.fudahospital.com/